CLINICAL TRIAL: NCT00896584
Title: May Pulseoximetry During Physical Exercise Predict Hypoxemia in COPD Patients During Air Travel?
Brief Title: Exercise Pulseoximetry for Pre-flight Evaluation of Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Type: Observational
Sponsor: LHL Helse (Other)
Responsible Party: Morten Ryg, Glittreklinikken
Other Study IDs: GK-40/3; S-08640b (REK); 2541 (Biobank); 2008/2/0079 (HelseRehab)
Record Dates: First submitted 2009-05-08; First posted 2009-05-11 (Estimated); Last update posted 2010-11-18 (Estimated); Status verified 2010-11

CONDITIONS: Chronic Obstructive Pulmonary Disease; Hypoxemia
Keywords: Chronic obstructive pulmonary disease; Hypoxemia; Pre-flight evaluation; Hypobaria; COPD; Pulseoximetry; Air travel; Exercise desaturation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypoxia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Some patients with chronic obstructive pulmonary disease (COPD) need supplementary oxygen during air travel. Guidelines issued by The British Thoracic Society (BTS) for pre-flight evaluation do not discriminate sufficiently between those who need supplementary oxygen during flight, and those who can do without. Previous studies have indicated that decreasing hemoglobin oxygen saturation during exercise may predict in-flight hypoxemia. The objective of the present study is to examine if adding exercise oxygen desaturation to the BTS algorithm will better predict requirements for in-flight supplementary oxygen.

DETAILED DESCRIPTION:
The British Thoracic Society (BTS) guidelines on pre-flight evaluation for patients with chronic respiratory disease is based on an algorithm where arterial oxygen saturation is the discriminating factor. It has recently been shown that this algorithm does not discriminate sufficiently between patients who need pre-flight evaluation and maybe supplementary oxygen during air travel, and those who can travel by air without supplemental oxygen or further evaluation. Studies have also shown that exercise desaturation may predict in-flight hypoxemia. The objective of the present study is to examine if inclusion of arterial oxygen saturation measured by pulseoximetry during exercise in the BTS algorithm, will increase the sensitivity and specificity of the BTS pre-flight evaluation guidelines.The study also include questionnaires on symptoms during air travel carried out before ande after the pre-flight evaluation.

ELIGIBILITY:
Inclusion Criteria:

* patients with COPD who have performed a hypoxia altitude simulation test
* able to perform the 6-minute walking test

Exclusion Criteria:

* unstable angina
* uncontrolled hypertension
* uncontrolled arrythmia
* patients with long-term oxygen treatment

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-05; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Edvardsen, MSc, Principal Investigator — LHL Helse; Morten S Ryg, Dr philos, Study Director — LHL Helse
Locations (1):
- Glittreklinikken, Hakadal, Hakadal, Norway

REFERENCES:
- [Background] Akero A, Christensen CC, Edvardsen A, Ryg M, Skjonsberg OH. Pulse oximetry in the preflight evaluation of patients with chronic obstructive pulmonary disease. Aviat Space Environ Med. 2008 May;79(5):518-24. doi: 10.3357/asem.2120.2008. PMID 18500050
- [Background] Akero A, Christensen CC, Edvardsen A, Skjonsberg OH. Hypoxaemia in chronic obstructive pulmonary disease patients during a commercial flight. Eur Respir J. 2005 Apr;25(4):725-30. doi: 10.1183/09031936.05.00093104. PMID 15802350
- [Background] British Thoracic Society Standards of Care Committee. Managing passengers with respiratory disease planning air travel: British Thoracic Society recommendations. Thorax. 2002 Apr;57(4):289-304. doi: 10.1136/thorax.57.4.289. No abstract available. PMID 11923546
- [Derived] Edvardsen A, Ryg M, Akero A, Christensen CC, Skjonsberg OH. COPD and air travel: does hypoxia-altitude simulation testing predict in-flight respiratory symptoms? Eur Respir J. 2013 Nov;42(5):1216-23. doi: 10.1183/09031936.00157112. Epub 2012 Dec 20. PMID 23258777